CLINICAL TRIAL: NCT04649307
Title: Cognitive Behavioral Therapy Following Myocardial Infarction
Acronym: MI-CBT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Brjann Ljotsson, Associate Professor, Karolinska Institutet
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MI-CBT
Record Dates: First submitted 2020-11-24; First posted 2020-12-02 (Actual); Last update posted 2022-05-24 (Actual); Status verified 2022-05

CONDITIONS: Myocardial Infarction
Keywords: CBT; Cardiac anxiety; Quality of Life; Physical activity
MeSH Terms: conditions — Myocardial Infarction; Motor Activity

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MI-CBT (Other): The treatment will be based on the AF treatment developed by the research group and further be developed and adapted during the course the study, based on the clinical presentation of the MI patients and their response to the CBT interventions detailed below. The MI-specific CBT will consist of 8 weekly face-to face digital video sessions with home assignments that can be reviewed and reported in the research groups secure platform. CBT for MI primarily targets two processes of disability; cardiac anxiety, and depressive inactivity
  Interventions: Behavioral: MI-CBT

INTERVENTIONS:
Behavioral: MI-CBT — Education, Interoceptive exposure, Exposure in-vivo, Behavioral activation, Relapse prevention

SUMMARY:
Myocardial infarction (MI) is one of the leading cause s of health loss globally, representing a large proportion of general disability. Anxiety and depression occur in 20-30 percent of patients following MI and have been identified as risk factors for recurrent adverse cardiac event. The purpose of our this study is to develop and evaluate a disease specific cognitive behavioral therapy (C BT) protocol to reduce cardia anxiety, depression, increase physical inactivity and quality of life (Q oL) in patients following MI.

DETAILED DESCRIPTION:
The study will include 20 patients. The MI-specific CBT lasts for 8 weeks and is delivered face-to-face via a secure digital video solution (to minimize cancelled sessions because of the COVID-19 pandemic) or at the Karolinska Universitetssjukhuset cardiac research unit, by licensed psychologists with expertise in CBT for cardiac disease. During treatment, the psychologists will have direct access to a cardiologist assigned to the project and treatments are conducted in close interdisciplinary collaboration to ensure patient safety.

ELIGIBILITY:
Inclusion Criteria:

( - )MI ≥ 6 months before assessment (type 1 STEMI/NSTEMI) ( - )Age 18-69 years endorsed cardiac anxiety that leads to significant distress or interferes with daily life (Cardiac Anxiety Questionnaire (CAQ); score ≥20) ( - ) On optimal medical treatment ( - )Able to read and write in Swedish.

Exclusion Criteria:

( - ) heart failure with severe systolic dysfunction (ejection fraction ≤ 35%) ( - ) significant valvular disease ( - ) planned coronary artery bypass surgery or other invasive therapy ( - ) other severe medical illness ( - )any medical restriction to physical exercise ( - )severe psychiatric disorder, severe depression, or risk of suicide ( - )alcohol dependency.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2020-12-29 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2021-12-01 (Actual)

PRIMARY OUTCOMES:
Cardiac anxiety questionnaire | baseline
  Measure of cardiac anxiety, fear, avoidance and attention. The score ranges between 0 and 72, with a greater score indicating elevated cardiac anxiety.
Cardiac anxiety questionnaire | 2 months from baseline
  Measure of cardiac anxiety, fear, avoidance and attention. The score ranges between 0 and 72, with a greater score indicating elevated cardiac anxiety.
Cardiac anxiety questionnaire | 8 months from baseline
  Measure of cardiac anxiety, fear, avoidance and attention. The score ranges between 0 and 72, with a greater score indicating elevated cardiac anxiety.

SECONDARY OUTCOMES:
12-Item Short-Form Health Survey (SF-12) | Baseline
  General quality of life, with a score ranging from 0 to 100. A higher score indicating a better quality of life.
12-Item Short-Form Health Survey (SF-12) | 2 months from baseline
  General quality of life, with a score ranging from 0 to 100. A higher score indicating a better quality of life.
12-Item Short-Form Health Survey (SF-12) | 8 months from baseline
  General quality of life, with a score ranging from 0 to 100. A higher score indicating a better quality of life.
Body Sensation Questionnaire | Baseline
  Fear of bodily symptoms, score ranging from 0 to 72 . Higher scores indicate more fear of body sensations.
Body Sensation Questionnaire | 2 months from baseline
  Fear of bodily symptoms, score ranging from 0 to 72 . Higher scores indicate more fear of body sensations.
Body Sensation Questionnaire | 8 months from baseline
  Fear of bodily symptoms, score ranging from 0 to 72 . Higher scores indicate more fear of body sensations.
Patient Health Questionnaire-9 | Baseline
  Measure of depression, score ranging 0 to 27 with a higher score indicating higher level of depression.
Patient Health Questionnaire-9 | 2 months from Baseline
  Measure of depression, score ranging 0 to 27 with a higher score indicating higher level of depression.
Patient Health Questionnaire-9 | 8 months from Baseline
  Measure of depression, score ranging 0 to 27 with a higher score indicating higher level of depression.
Generalized Anxiety Disorder 7-item | Baseline
  General anxiety, score ranging from 0-21, with a higher score indicating more anxiety and worry.
Generalized Anxiety Disorder 7-item | 2 months from baseline
  General anxiety, score ranging from 0-21, with a higher score indicating more anxiety and worry.
Generalized Anxiety Disorder 7-item | 8 months from baseline
  General anxiety, score ranging from 0-21, with a higher score indicating more anxiety and worry.
The Godin Leisure-time Exercise | Baseline
  Level of physical activity. The participant rate numbers of time per week that they engage in physical activity. The numb ers are the categorized in to low, moderate, and high levels of physical activity.
The Godin Leisure-time Exercise | 2 months from Baseline
  Level of physical activity. The participant rate numbers of time per week that they engage in physical activity. The numb ers are the categorized in to low, moderate, and high levels of physical activity.
The Godin Leisure-time Exercise | 8 months from Baseline
  Level of physical activity. The participant rate numbers of time per week that they engage in physical activity. The numb ers are the categorized in to low, moderate, and high levels of physical activity.
Tampas Scale for Kinesophobia-Heart version | Baseline
  Fear of physical activity. The total score varies between 17 and 68, with higher values indicating more severe kinesiophobia.
Tampas Scale for Kinesophobia-Heart version | 2 months from Baseline
  Fear of physical activity. The total score varies between 17 and 68, with higher values indicating more severe kinesiophobia.
Tampas Scale for Kinesophobia-Heart version | 8 months form Baseline
  Fear of physical activity. The total score varies between 17 and 68, with higher values indicating more severe kinesiophobia.
Client satisfaction Questionnaire | 2 months from Baseline
  Treatment satisfaction, score ranging from 0 to 32, with a higher score indication more satisfaction with the treatment.
Adverse events | 2 months from baseline
  Potential adverse reactions to the treatment. Participants will be asked to report and rate the short- and long term discomfort of the adverse event on a scale from 0 ('did not affect me at all') and 3 ('affected me very negatively').
Adverse events | 8 months from baseline
  Potential adverse reactions to the treatment. Participants will be asked to report and rate the short- and long term discomfort of the adverse event on a scale from 0 ('did not affect me at all') and 3 ('affected me very negatively').

CONTACTS AND LOCATIONS:
Locations (1):
- Karolinska University Hospital, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No